CLINICAL TRIAL: NCT05685277
Title: Open-label With Blinding Bioanalytical Stage Randomized Crossover Two Period Two Sequences Single Dose Bioequivalence Study of Two Formulations Ramipril/Hydrochlorothiazide Tablets 10 mg/25 mg (Manufacturer: Pharmtechnology LLC, Republic of Belarus) and Tritace® Plus Tablets 10 mg/25 mg (Manufacturer: Sanofi S.p.A., Italy; Holder of the Registration Certificate: Sanofi-Aventis Deutschland GmbH, Germany) in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Two Formulations of Tablets Ramipril/Hydrochlorothiazide 10 mg/25 mg in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Ligand Research, LLC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RMPL-HCTZ-2021
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-08

CONDITIONS: Bioequivalence
Keywords: Ramipril; Hydrochlorothiazide; Bioequivalence; Tritace® Plus
MeSH Terms: interventions — Ramipril; Hydrochlorothiazide; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence TR (Other): 25 subjects assigned to the sequence TR will receive a single 10 mg/25 mg dose of the test product Ramipril/Hydrochlorothiazide (1 x 10 mg/25 mg tablet), marked as T in the sequence, in Period 1 and a single 10 mg/25 mg dose of the reference product Tritace® Plus (1 x 10 mg/25 mg tablet), marked as R in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Ramipril/Hydrochlorothiazide tablet 10 mg/25 mg; Drug: Tritace® Plus tablet 10 mg/25 mg
- Sequence RT (Other): 25 subjects assigned to the sequence RT will receive a single 10 mg/25 mg dose of the test product Tritace® Plus (1 x 10 mg/25 mg tablet), marked as R in the sequence, in Period 1 and a single 10 mg/25 mg dose of the reference product Ramipril/Hydrochlorothiazide (1 x 10 mg/25 mg tablet), marked as T in the sequence, in period 2. These treatments will be administered orally with approximately 200 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Ramipril/Hydrochlorothiazide tablet 10 mg/25 mg; Drug: Tritace® Plus tablet 10 mg/25 mg

INTERVENTIONS:
Drug: Ramipril/Hydrochlorothiazide tablet 10 mg/25 mg — Ramipril/Hydrochlorothiazide is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 10 mg of ramipril and 25 mg of hydrochlorothiazide.
  Other Names: The test product
Drug: Tritace® Plus tablet 10 mg/25 mg — Tritace® Plus is manufactured by Sanofi S.p.A., Italy (holder of the registration certificate: Sanofi-Aventis Deutschland GmbH, Germany). Each tablet contains 10 mg of ramipril and 25 mg of hydrochlorothiazide.
  Other Names: The reference product

SUMMARY:
This is an open-labeled, with blinding bioanalytical stage, randomized, two period, two sequences, single-center, crossover, comparative study, where each participant will be randomly assigned to the reference (Tritace® Plus, 10 mg/25 mg tablets) or the test (Ramipril/Hydrochlorothiazide, 10 mg/25 mg tablets) formulation in each period of study (sequences Test-Reference (TR) or Reference-Test (RT)), in order to evaluate if both formulations are bioequivalent.

DETAILED DESCRIPTION:
This is an open-labeled, with blinding bioanalytical stage, randomized, two period, crossover, a single-center, comparative, single-dose study, in which 50 healthy adult subjects will receive one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of combination ramipril/hydrochlorothiazide after a single oral dose administration under fasting conditions.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 12 hours prior to drug administration for each study period.

Hospitalization in the first period of the study will last no more than 36 hours, after which, in the absence of indications for an extension of hospitalization, each subject will be released home; after that, the first period of the study will be completed.

The procedures of the second study period will be identical to the first period.

After completing all the procedures of the second study period, each subject will undergo a final examination, after which, in case of the absence of adverse events and indications for prolonging hospitalization, the study for the subjects will be considered completed.

The total duration of the study for the subject will be no more than 46 days.

Eligible subjects will be randomized to one of two treatment sequences. There will be two sequences in the study: TR and RT, where T = the test product, R = the reference product.

For each study period, subjects will receive a single 10 mg/25 mg oral dose of ramipril/hydrochlorothiazide (the test or the reference formulation). Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Fasting will continue for at least 4 hours following drug administration. Breakfast will be organized 4 hours after taking the drug, lunch after 8 hours, dinner after 12 hours.

Water will be provided as needed until 1 hour predose. Water will be allowed beginning 2 hours after the administration of the drug.

A total of 24 blood samples will be collected (one tube of 6 mL each) in each study period for pharmacokinetic (PK) assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 72 hours after drug administration.

The concentration of ramipril, ramiprilat and hydrochlorothiazide will be determined using high performance liquid chromatography with mass spectrometric detection according to a method developed and validated in the analytical laboratory.

Statistical analysis of all PK parameters will be based on an ANOVA model. Two-sided 90% confidence interval of the ratio of geometric LSmeans obtained from the ln-transformed PK parameters will be calculated.

Statistical inference of ramipril, ramiprilat and hydrochlorothiazide will be based on a bioequivalence approach using the following standards: the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and the Reference for the ln-transformed parameters Cmax and AUC0-72 should all be within the 80.00 to 125.00% bioequivalence range.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women aged between 18 to 45 years, inclusive;
2. Body mass index 18.5-30.0 kg/m², inclusive;
3. Verified diagnosis "healthy" according to the standard clinical, laboratory and instrumental examination methods;
4. The level of systolic blood pressure (SBP) ≥100 mm Hg and ≤ 130 mm Hg and diastolic blood pressure (DBP) ≥ 70 mm Hg and ≤ 90 mm Hg; heart rate more than 60 beats/min and less than 90 beats/min at the time of screening, respiratory rate more than 12 and less than 20 per minute at the time of screening, body temperature above 35.9 ° C and below 36.9 °C at the time of screening;
5. Subjects are able to understand the requirements of the study;
6. Subjects are able to accept all the restrictions imposed during the course of the study;
7. Availability of written informed consent of the volunteer to participate in the study in accordance with applicable law, obtained before the start of any research procedures;
8. For female subject with preserved reproductive potential: negative pregnancy test and consent to use adequate methods of contraception from the first day of screening up to 30 days after taking the drug in the second period, or the absence of reproductive potential; in the case of using hormonal contraceptives, they must be canceled at least 2 months before the first day of screening;
9. For male: consent to use adequate methods of contraception with partners with preserved reproductive potential from the first day of screening up to 30 days after taking the drug in the second period.

Exclusion Criteria:

1. Drug intolerance to any drug;
2. Burdened allergic history;
3. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption;
4. Acute infectious diseases or allergic reactions requiring treatment (including drug allergies) less than 4 weeks before the first day of screening;
5. Surgical interventions on the gastrointestinal tract, with the exception of appendectomy;
6. Volunteers with suspected hypersensitivity to study drugs or any of their components;
7. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood or other conditions that make it impossible for a volunteer to participate in the study according to the opinion of the researcher;
8. The value of standard laboratory and instrumental parameters that go beyond the reference values;
9. Positive test for syphilis, hepatitis B, hepatitis C, HIV or nasal and oropharyngeal swab for SARS-CoV-2;
10. Positive test for alcohol in exhaled air;
11. Positive urine analysis for the content of narcotic and potent substances;
12. For women - positive pregnancy test;
13. Any diet, such as vegetarian, within 2 weeks prior to the first day of screening;
14. Intake of more than 10 units alcohol per week (1 unit of alcohol is equivalent to 500 ml of beer, 200 ml of wine or 50 ml of spirits ethyl 40%) or history of alcoholism, drug addiction, drug abuse;
15. Inability to go without food for at least 12 hours and the inability to take the drug on an empty stomach;
16. Donation of plasma or blood (450 ml or more) less than 3 months before the first day of screening;
17. Depot injections, installation of intrauterine hormonal therapeutic systems or implants of any drugs 6 months before the first day of screening;
18. For women: use of hormonal contraceptives less than 2 months before the first day of screening;
19. Regular medication intake less than 2 weeks before the first day of screening;
20. Taking drugs that have a pronounced effect on hemodynamics, liver function, etc. (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants, tagamet, cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones , antihistamines), vitamins, dietary supplements, herbal preparations, including cat's claw, medicinal angelica, evening primrose, feverfew, garlic, ginger, ginkgo, red clover, horse chestnut, green tea, ginseng; Hypericum perforatum, etc. less than 30 days before the first day of screening;
21. For women: volunteers with saved reproductive potential who had unprotected intercourse with an unsterilized male partner within 30 days prior to the first day of screening;
22. For women: the period of breastfeeding;
23. Participation in any other clinical trial or use of investigational drugs less than 3 months prior to the first day of screening;
24. Difficult access to the vein, complicating or making it impossible to install a catheter and frequent blood sampling;
25. Smoking;
26. Volunteers who are unwilling or unable to give up alcohol and excessive physical activity from the first day of screening until the follow-up visit;
27. Volunteers who are unwilling or unable to avoid drinks and foods containing methylxanthines and grapefruit/grapefruit juice, as well as foods containing poppy from the first day of screening until the follow-up visit;
28. Volunteers who lead a lifestyle (including night work and extreme physical activity such as sports or heavy lifting) that may make it difficult to interpret the laboratory data obtained during the study;
29. Volunteers who do not intend to comply with the study regime and / or do not inspire confidence in the researcher;
30. Volunteers who are obviously or likely, in the opinion of the investigator, unable to understand and evaluate the information on this study as part of the process of signing the informed consent form, in particular regarding the expected risks and possible discomfort;

29. Dehydration due to diarrhea, vomiting or other reason within the last 24 hours prior to the first day of screening; 30. The presence of seizures, epilepsy and any other neurological disorders in the history of volunteers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Cmax of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Maximum observed concentration in plasma.
AUC0-72 of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) at the 72 hour time point using the linear trapezoidal method.

SECONDARY OUTCOMES:
Tmax of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value.
TLQC of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Time of last observed quantifiable concentration.
AUC0-INF of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant).
Residual area of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Extrapolated area (i.e. percentage of AUC0-INF due to extrapolation from TLQC to infinity).
Time point where the log-linear elimination phase begins (TLIN) of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Time point where the log-linear elimination phase begins.
λZ of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve.
Terminal elimination half-life (Thalf) of ramipril, ramiprilat and hydrochlorothiazide in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ.
Number of treatment-emergent adverse events for the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.10, 0.20, 0.30, 0.45, 1.00, 1.15, 1.30, 1.45, 2.00, 2.30, 3.00, 3.30, 4.00, 4.30, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 24.00, 48.00, 72.00 hours after each drug administration.
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Filatov, Study Director — Ligand Research, LLC; Irina Rodyukova, Principal Investigator — Ligand Research, LLC
Locations (1):
- Separate medical division "Comed" (Ligand Research LLC), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No